CLINICAL TRIAL: NCT01462890
Title: A Prospective Randomised Phase III Trial to Evaluate Optimal Treatment Duration of First-line Bevacizumab in Combination With Carboplatin and Paclitaxel in Patients With Primary Epithelial Ovarian, Fallopian Tube or Peritoneal Cancer
Brief Title: Evaluation of Optimal Treatment Duration of Bevacizumab Combination With Standard Chemotherapy in Patients With Ovarian Cancer
Acronym: BOOST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Study Group (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other); Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 17
Record Dates: First submitted 2011-10-25; First posted 2011-11-01 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Genital Diseases, Female; Ovarian Diseases; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: Ovarian Carcinoma; Bevacizumab; Paclitaxel; Carboplatin
MeSH Terms: conditions — Genital Diseases, Female; Ovarian Diseases; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Randomized Phase III study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Other): Patients receive bevacizumab iv followed by paclitaxel iv and carboplatin iv on day 1. Treatment repeats every 3 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then continue to receive bevacizumab iv alone every 3 weeks for 16 cycles.
  Interventions: Biological: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin; Other: specialized pathology review (Germany only)
- Research Arm (Experimental): Patients receive bevacizumab iv followed by paclitaxel iv and carboplatin iv on day 1. Treatment repeats every 3 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then continue to receive bevacizumab iv alone every 3 weeks for 38 cycles.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Other: specialized pathology review (Germany only)

INTERVENTIONS:
Biological: Bevacizumab — 15 mg/kg, iv on day 1 every 3 weeks up to and including cycle 22 vs cycle 44
  Arms: Control Arm
Drug: Paclitaxel — 175 mg/m², iv on day 1 every 3 weeks for 6 cycles
Drug: Carboplatin — AUC 5, iv on day 1 every 3 weeks for 6 cycles
Other: specialized pathology review (Germany only) — before randomization

SUMMARY:
The purpose of this study is to determine whether the early and continuous addition of bevacizumab for up to 30 months to the standard chemotherapy is more effective than the early and continuous addition of bevacizumab for up to 15 months.

DETAILED DESCRIPTION:
Determination whether the early and continuous addition of bevacizumab for up to 30 months to the standard chemotherapy is more effective than the early and continuous addition of bevacizumab for up to 15 months

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to initiation of any study specific procedures and treatment as confirmation of the patients awareness and willingness to comply with the study requirements
* Primary diagnosis is confirmed by specialized pathology review (Germany only)
* Females aged ≥ 18 years
* Histologically confirmed, newly diagnosed

  * Epithelial ovarian carcinoma
  * Fallopian tube carcinoma
  * Primary peritoneal carcinoma AND FIGO stage IIb - IV (all grades and all histological types)
* Patients should have already undergone surgical debulking, by a surgeon experienced in the management of ovarian cancer, with the aim of maximal surgical cytoreduction according to the GCIG Conference Consensus Statement. There must be no planned surgical debulking prior to disease progression. Patients with stage III and IV disease in whom initial surgical debulking was not appropriate or possible will still be eligible providing

  * the patient has a histological diagnosis and
  * debulking surgery prior to disease progression is not foreseen
* Patients must be able to commence cytotoxic chemotherapy within 8 weeks of cytoreductive surgery. The first dose of bevacizumab can be omitted in both arms if the investigator decides to start chemotherapy within 4 weeks of surgery.
* ECOG 0-2
* Life expectancy > 3 months
* Adequate bone marrow function (within 14 days prior to randomization)

  * ANC ≥ 1.5 x 10^9/L
  * PLT ≥ 100 x 10^9/L
  * Hb ≥ 9 g/dL (can be post-transfusion)
* Adequate coagulation parameters (within 14 days prior to randomization)

  * Patients not receiving anticoagulant medication who have an INR ≤ 1.5 and an aPTT ≤ 1.5 x ULN
  * The use of full-dose oral or par-enteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to institution medical standard) and the patient has been on a stable dose of anticoagulants for at least two weeks at the time of randomization.
* Adequate liver function (within 14 days prior to randomization)

  * Serum bilirubin ≤ 1.5 x ULN
  * Serum transaminases ≤ 2.5 x ULN
* Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2+, 24 hour urine must demonstrate ≤ 1 g of protein in 24 hours
* Adequate postoperative GFR > 40 ml/min (estimates based on the Cockroft-Gault or Jelliffe formula are sufficient)

Exclusion Criteria:

* Non-epithelial origin of the ovary, the fallopian tube or the peritoneum
* Borderline tumours (tumours of low malignant potential) and FIGO stage Ia - IIa tumours
* Planned intraperitoneal cytotoxic chemotherapy
* Prior systemic anti-cancer therapy for ovarian cancer (for example chemotherapy, monoclonal antibody therapy, tyrosine kinase inhibitor therapy or hormonal therapy)
* Surgery (including open biopsy) within 4 weeks prior to anticipated first dose of bevacizumab (allowing for the fact that bevacizumab can be omitted from the first cycle of chemotherapy). It is strongly recommended that an interval of 7 days is left between the insertion of any central venous access devices (CVADs) and the onset of bevacizumab treatment.
* Any planned surgery during the study treatment period plus 4 additional weeks to allow for bevacizumab clearance
* Uncontrolled hypertension (sustained elevation of BP systolic > 150mmHg and/or diastolic > 100mmHg despite antihypertensive therapy)
* Any previous radiotherapy to the abdomen or pelvis
* Significant traumatic injury during 4 weeks preceding the potential first dose of bevacizumab
* History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to randomization) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to randomization) in case of suspected spinal cord compression.
* History or evidence upon neurological examination of central nervous system (CNS) disease, unless adequately treated with standard medical therapy e.g. uncontrolled seizures
* Previous Cerebro-Vascular Accident (CVA), Transient Ischaemic Attack (TIA) or Sub-Arachnoid Haemorrhage (SAH) within 6 months prior to randomization
* Fertile woman of childbearing potential not willing to use adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) for the study duration and at least 6 months afterwards
* Pregnant or lactating women
* Treatment with other investigational agents, or participation in another clinical trial testing a drug within the past 4 weeks before start of therapy concomitantly with this trial
* Malignancies other than ovarian cancer within 5 years prior to randomization, except for adequately treated

  * carcinoma in situ of the cervix
  * and/or basal cell skin cancer
  * and/or non-melanomatous skin cancer
  * carcinoma in situ of the breast
  * and/or early endometrial carcinoma as specified below. Patients may have received previous adjuvant chemotherapy for other malignancies e.g. breast or colorectal carcinoma if diagnosed over 5 years ago with no evidence of subsequent recurrence.
* Patients with synchronous primary endometrial carcinoma, or a past history of primary endometrial carcinoma, are excluded unless ALL of the following criteria for describing the endometrial carcinoma are met

  * Disease stage FIGO stage ≤ IA (tumour invades less than one half of the myometrium)
* Known hypersensitivity to bevacizumab and its excipients, Chinese hamster ovary cell products or other recombinant human or humanised antibodies
* Non healing wound, active ulcer or bone fracture. Patients with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection are eligible but require 3 weekly wound examinations
* History or evidence of thrombotic or hemorrhagic disorders within 6 months prior to randomization
* Clinically significant cardiovascular disease, including

  * Myocardial infarction or unstable angina within 6 months of randomization
  * NYHA ≥ Grade 2 Congestive Heart Failure (CHF)
  * Poorly controlled cardiac arrhythmia despite medication (patients with rate-controlled atrial fibrillation are eligible)
  * Grade ≥ 3 peripheral vascular disease (i.e. symptomatic and interfering with activities of daily living requiring repair or revision)
* Current or recent (within 10 days prior to randomization) chronic use of aspirin > 325 mg/day
* Pre-existing sensory or motor neuropathy ≥ Grade 2
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicates the use of an investigational drug or puts the patient at high risk for treatment-related complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | every 12 weeks until progression or up to 30 months, thereafter every 6 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | every 12 weeks until progression or up to 30 months, thereafter every 6 months
Overall survival (OS) | every 3 weeks, 31 months after start of treatment, thereafter every 6 months
Health related Quality of life (QoL) | baseline, then every 12 weeks until progression, 31 months after start of treatment or if applicable 4 weeks after last dose of bevacizumab (whichever occurs later)
Safety and tolerability, i.e. type, frequency, severity and duration of adverse reactions | every 3 weeks, 31 months after start of treatment or if applicable 4 weeks after last dose of bevacizumab (whichever occurs later)
Translational Research - Tumor Tissue Block | Assessment at end of study planned
  may be obtained at any time during therapy, preferably at cycle 1 or at a subsequent visit
Translational Research - Complementary and Alternative Treatment Questionnaires | baseline, 6 months and 12 months after start of treatment, if required at timepoint of treatment termination

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Pfisterer, MD PhD, Study Chair — AGO Study Group
Locations (131):
- Denmark (3):
  - Aalborg
  - Copenhagen
  - Herlev
- Finland (4):
  - Kuopio
  - Oulu
  - Tampere
  - Turku
- France (33):
  - Angers
  - Besançon
  - Blois
  - Bordeaux
  - Caen
  - Cahors
  - Clamart
  - Clermont-Ferrand
  - Créteil
  - Dax
  - Draguignan
  - Grenoble
  - Limoges
  - Lyon
  - Mougins
  - Nancy
  - Nantes
  - Nice
  - Nîmes
  - Orléans
  - Paris
  - Pau
  - Plérin
  - Poitiers
  - Quimper
  - Reims
  - Rouen
  - Saint-Herblain
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Vannes
  - Villejuif
- Germany (86):
  - Aachen
  - Arnsberg
  - Aschaffenburg
  - Augsburg
  - Bad Homburg
  - Berlin
  - Bochum
  - Bonn
  - Bottrop
  - Brandenburg
  - Bremen
  - Chemnitz
  - Coburg
  - Cologne
  - Deggendorf
  - Dessau
  - Dresden
  - Düsseldorf
  - Ebersberg
  - Eggenfelden
  - Erlangen
  - Essen
  - Esslingen am Neckar
  - Flensburg
  - Frankfurt/M.
  - Freiburg im Breisgau
  - Fürstenfeldbruck
  - Fürth
  - Georgsmarienhütte
  - Gera
  - Göttingen
  - Greifswald
  - Gütersloh
  - Halle
  - Hamburg
  - Hanau
  - Hanover
  - Heidelberg
  - Henstedt-Ulzburg
  - Hildesheim
  - Jena
  - Kaiserslautern
  - Karlsruhe
  - Kassel
  - Kiel
  - Krefeld
  - Lich
  - Limburg
  - Lübeck
  - Lüneburg
  - Magdeburg
  - Mainz
  - Mannheim
  - Marburg
  - Minden
  - München
  - Neumarkt
  - Neuss
  - Nordhausen
  - Offenbach
  - Offenburg
  - Oldenburg
  - Osnabrück
  - Ravensburg
  - Regensburg
  - Reutlingen
  - Rosenheim
  - Rostock
  - Rottweil
  - Saalfeld
  - Salzgitter
  - Schwäbisch Hall
  - Schweinfurt
  - Sigmaringen
  - Solingen
  - Stralsund
  - Stuttgart
  - Torgau
  - Trier
  - Tübingen
  - Ulm
  - Viersen
  - Wiesbaden
  - Witten
  - Wolfsburg
  - Worms
- Norway (3):
  - Bergen
  - Oslo
  - Trondheim
- Sweden (2):
  - Falun
  - Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Pfisterer J, Joly F, Kristensen G, Rau J, Mahner S, Pautier P, El-Balat A, Kurtz JE, Canzler U, Sehouli J, Heubner ML, Hartkopf AD, Baumann K, Hasenburg A, Hanker LC, Belau A, Schmalfeldt B, Denschlag D, Park-Simon TW, Selle F, Jackisch C, Burges A, Luck HJ, Emons G, Meier W, Gropp-Meier M, Schroder W, de Gregorio N, Hilpert F, Harter P. Optimal Treatment Duration of Bevacizumab as Front-Line Therapy for Advanced Ovarian Cancer: AGO-OVAR 17 BOOST/GINECO OV118/ENGOT Ov-15 Open-Label Randomized Phase III Trial. J Clin Oncol. 2023 Feb 1;41(4):893-902. doi: 10.1200/JCO.22.01010. Epub 2022 Nov 4. PMID 36332161